CLINICAL TRIAL: NCT01884922
Title: PHASE I-II STUDY OF VINBLASTINE IN COMBINATION WITH NILOTINIB IN CHILDREN, ADOLESCENTS, AND YOUNG ADULTS WITH REFRACTORY OR RECURRENT LOW-GRADE GLIOMA
Brief Title: Study Of Vinblastine in Combination With Nilotinib in Children, Adolescents and Young Adults
Acronym: VINILO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-003005-10 Phase I; 2012/1883 (Other: CSET number); 022 (Other: ITCC)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Refractory Low-grade Gliomas; Recurrent Low-grade Gliomas
Keywords: Children; adolescents; young adults
MeSH Terms: interventions — nilotinib; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): Nilotinib (Tasigna®): 115 to 350 mg/m2 twice daily (BID) orally given continuously (115 mg/m2 once daily if de-escalation requested
  Vinblastine: 3 to 6 mg/m2 once weekly in a 15-minute infusion, on Days 1, 8, 15 and 22 of each cycle.
  Interventions: Drug: Nilotinib; Drug: Vinblastine

INTERVENTIONS:
Drug: Nilotinib — Tasigna®(nilotinib):: 50 mg, 150 mg and 200 mg capsules. Tasigna® capsules contain lactose monohydrate, crospovidone, poloxamer, colloidal silicon dioxide and magnesium. Orally; the capsules should be swallowed as a whole with water. No food should be consumed for 2 hours before the dose is taken and for at least one hour thereafter. For patients who are unable to swallow capsules, the content of each capsule may be dispersed in one teaspoon of apple sauce or compote or nonfat plain yogurt and should be taken immediately. Not more than one teaspoon of apple sauce / yogourt, and no food other than apple sauce or nonfat plain yogurt must be used.
  Other Names: Tasigna®
Drug: Vinblastine — Vinblastine: 3 to 6 mg/m2 once weekly in a 15-minute infusion, on Days 1, 8, 15 and 22 of each cycle.
  Each 28-day cycle is repeated on Day 29/Day 1. No intra-patient doseescalation is permitted. Dose allocation will be centrally defined, based on toxicity observed in patients previously evaluated. Every new patient will be treated at the best current recommended dose, i.e. the dose associated with an estimated level of toxicity that is judged acceptable (20% DLT). At least two patients fully observed with no DLT are requested at a given dose level before dose escalation.

SUMMARY:
Multicenter, open label, prospective study including successively a phase I trial and then a phase II trial Phase I : Open label, non-randomized, sequential dose escalation of both drugs, vinblastine and nilotinib.

DETAILED DESCRIPTION:
Low grade gliomas (LGG) are the most frequent brain tumor type in children. They are often chemosensitive. However, more than 50% of these tumors will progress within the first 5 years after the start of the treatment and need a second-line therapy (Laithier, JCO 2003). In most cases, patients are still young and the risk of side effects from radiation therapy will call for another medical treatment. If a tumor does not respond to first-line chemotherapy, the prognosis worsens with 25% of deaths within the first 5 years for optic gliomas (de Haas, Pediatr Blood Cancer 2009). Vinblastine (Velbe®) is an effective drug for low grade gliomas with both antiproliferative and antiangiogenic effects. An update of the Canadian phase II of weekly vinblastine (6 mg/m²/week) reported one complete response (CR), three partial responses (PR) and 9 minor responses (MR) in the first 31 patients (Bouffet, Abstract in Neuro-Oncology 2008). The 1-year progressionfree survival (PFS) rate was 57%. Tolerance of the treatment is fair allowing prolonged maintenance therapy as in Langerhans cell histiocytosis and anaplastic large cell lymphoma (ALCL). These data encourage proceeding with further testing this approach in pediatric low-grade glioma.

Nilotinib is a tyrosine kinase inhibitor (TKI) known to affect c-Kit, DDR1 and the PDGF receptors alpha and beta. PDGF is a growth factor for normal and tumoral astrocytes and oligodendrocytes. In addition, PDGF receptors are expressed on pediatric low-grade glioma vessels (McLaughlin, J Pediatr Hematol Oncol 2003; Peyrl, Pediatr Blood Cancer 2009). Tumor response to this class of TKI has been reported occasionally (Peyrl, Pediatr Blood Cancer 2009; McLaughlin, J Pediatr Hematol Oncol 2003). When used as monotherapy, this class of TKI was well tolerated in children, including those with brain tumors (Wayne, Blood 2008; Baruchel, Eur J Cancer 2009; Geoerger, Eur J Cancer 2009). Taking advantage of their different antiangiogenic mechanisms, their limited and non-overlapping toxicities, vinblastine and nilotinib could play an interesting role in the treatment of pediatric low-grade glioma. Nilotinib via PDGFRA and c-kit interactions may also interfere with the stroma of the tumor which is a key factor for tumor growth as shown in the NF1 mouse model (Daginakatte, Cancer Res 2008; Kim, Neuroscience 2010; Simmons, J Neuropathol Exp Neurol 2011). Both drugs have also immunostimulating effects especially in dendritic cells, that will be explored during treatment in selected patients (Tanaka, Cancer Res 2009; Nishioka Immunotherapy 2011) Previous to the phase II assessing the efficacy of the combination compared to vinblastine as single agent, nilotinib and vinblastine have to be administered by escalating dosages in order to identify the recommended doses of each agent when given in combination. This phase I part of the trial is justified by a possible interaction of the two drugs that are substrates of cytochrome P450 CYP3A4. Initial/starting dose of nilotinib (115 mg/m² BID) will be 50% of the recommended dose when used as monotherapy in adults (800 mg/day: 400 mg BID =230 mg/m2 BID). Initial/starting dose of vinblastine will be 50% of the recommended dose when used as monotherapy or in association with other chemotherapeutic drugs (i.e. 3 mg/m2 once a week). This justifies obtaining pharmacokinetic data on both drugs when used in combination. A phase I trial evaluating nilotinib as single agent in pediatrics in hematological malignancies is ongoing, run by the ITCC and the COG group, exploring the dose-levels 230 mg/m² to 460 mg/m² BID. The results of this phase I trial, expected by 2012, and the data of the current trial will be considered to decide whether a higher dose-level for nilotinib can be opened (350 mg/m² BID).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed by the patient, or parents or legal representative and assent of the minor child.
2. Age: 6 months to < 21 years of age at time of study entry
3. Histologically confirmed low-grade glioma in non-NF1 patients (no further biopsy is needed at study entry). For patients with NF1 and optic pathway glioma, no biopsy is required to confirm the radiological diagnosis of the low grade glioma.
4. Relapse or refractory tumor after at least one first-line therapy, not taking into account surgery only.
5. Evaluable Disease on morphologic MRI
6. Karnofsky performance status score >=70% for patients >12 years of age, or Lansky score >=70% for patients <=12 years of age, including patients with motor paresis due to disease.
7. Administration of stable dose of steroids for at least one week
8. Life expectancy >= 3 months.
9. Adequate organ function:

   * Adequate hematopoietic function: neutrophils ³1.0 x 109/L, platelets ³100 x 109/L; hemoglobin ³8 g/dL
   * Adequate renal function: serum creatinine < 1.5 x ULN for age In others cases where serum creatinine >1.5 ULN according to age, Glomerular filtration rate or creatinine clearance has to be >70 mL/min/1.73 m2 or >70% of the expected value
   * Adequate electrolytes levels: potassium, magnesium, phosphor, total calcium Lower Limit of Normal (LLN)
   * Adequate hepatic function: total bilirubin <=1.5 x ULN; AST and ALT <=2.5 x ULN.
   * Absence of peripheral neuropathy >= grade 2 (Common Toxicity Criteria Adverse Event, NCI CTCAE v4.0)
   * Adequate cardiac function:

   Shortening Fraction (SF) >= 28% (35% for children <3 years) and Left Ventricular Ejection Fraction (LVEF) >= 50% at baseline, as determined by echocardiography

   Absence of QTc prolongation (QTc > 450 msec on baseline ECG, using the QTcF formula) or other clinically significant ventricular or atrial arrhythmia
10. Wash-out period of at least

    * 3 weeks in case of preliminary chemotherapy,
    * 6 weeks in case of nitrosourea-containing chemotherapy,
    * 2 weeks in the case of treatment with vincristine only
    * 6 weeks in case of radiation therapy
11. Possibility of receiving the therapeutic schedule as indicated in the protocol
12. Patients with reproductive potential must use effective contraception during their treatment and for up to 90 days after the last dose. Females with reproductive potential must have a negative pregnancy test <= 7 days before starting Nilotinib and/or Vinblastine.
13. Patients already treated with one of the two drugs can be enrolled in the trial provided that rechallenging them with the same drug could be considered acceptable

Exclusion Criteria:

1. Concomitant anti-tumor treatment
2. Not recovered to <Grade 2 from the acute toxic effects of all prior chemotherapy, immunotherapy or radiotherapy
3. Known intolerance or hypersensitivity to Vinblastine
4. Existence of another severe systemic disease
5. Uncontrolled infections not responsive to antibiotics, antiviral medicines, or antifungal medicines,
6. Any concurrent illness which in the opinion of the investigator may interfere with the treatment and evaluation of the patient
7. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of nilotinib.
8. Simultaneous treatment with strong cytochromes P450 CYP3A4 inhibitors (e.g. antiepileptic drugs, see complete list in the Appendix 5).
9. Simultaneous treatment with antiarrythmic drugs and other drugs known to prolong QT interval (cloroquine, halofantrine, clarithromycin, haloperidol, methadone, moxifloxacin, bepridil, cisapride and pimozide). A list of QT prolonging compounds can be found at http://www.azcert.org/medical-pros/druglists/drug-lists.cfm (Appendix 6)
10. Impaired cardiac function including any one of the following:

    * Clinically significant resting brachycardia (<50 beats per minute).
    * QTc > 450 msec on baseline ECG. If QTc >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc.
    * Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension).
    * History of or presence of clinically significant ventricular or atrial tachyarrhythmias (including congenital long QT syndrome or a known family history of congenital long QT syndrome)

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
Safety Assessment - Dose-Limiting Toxicity (DLT) | Assessed over the first 28-day cycle
  Dose-Limiting Toxicity (DLT), assessed over the first 28-day cycle, defined as
  * Grade > 3 neutropenia (<1 x 109/L) for more than 7 days;
  * Grade > 2 thrombopenia (<75 x 109/L) or thrombocytopenia requiring transfusions for more than 7 days.
  * Grade 3 or grade 4 non-hematological toxicity, excluding grade 3 nausea, vomiting, fever, and hepatic toxicity that is rapidly reversible (i.e. returns to < 2.5 x ULN within 2 weeks after study drug discontinuation), and symptoms that are related to tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques GRILL, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (8):
- Medical University of Vienna, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- Gustave Roussy, Villejuif, Val De Marne, France
- University Hospital of Padua, Padua, Italy
- Erasmus MC/Sophia Children's Hospital, Rotterdam, Netherlands
- Fundació Sant Joan de Déu, Barcelona, Spain
- Swiss Pediatric Oncology Group, Bern, Switzerland
- Cancer Research UK Clinical Trials Unit School of Cancer Sciences University of Birmingham, Edgbaston, Birmingham, United Kingdom

REFERENCES:
- [Derived] Vairy S, Le Teuff G, Bautista F, De Carli E, Bertozzi AI, Pagnier A, Fouyssac F, Nysom K, Aerts I, Leblond P, Millot F, Berger C, Canale S, Paci A, Poinsignon V, Chevance A, Ezzalfani M, Vidaud D, Di Giannatale A, Hladun-Alvaro R, Petit FM, Vassal G, Geoerger B, Le Deley MC, Grill J. Phase I study of vinblastine in combination with nilotinib in children, adolescents, and young adults with refractory or recurrent low-grade glioma. Neurooncol Adv. 2020 Jun 9;2(1):vdaa075. doi: 10.1093/noajnl/vdaa075. eCollection 2020 Jan-Dec. PMID 32666050